CLINICAL TRIAL: NCT01729910
Title: Primary Care Child Obesity Intervention Targeting Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Tennessee State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R15HD054950-01A2 REVISED; 1R15HD054950-01A2 (NIH)
Record Dates: First submitted 2012-11-15; First posted 2012-11-20 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Overweight; Obesity
Keywords: overweight; obesity; rural; primary care
MeSH Terms: conditions — Overweight; Obesity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent education / behavioral counseling (Experimental): Parents of children in the intervention group will be invited to participate in four group visits and two individual visits with their primary care provider as well as four follow-up phone calls with study personnel (project coordinator or registered dietician). Providers and study personnel will be trained in the use of the NIH We Can! curriculum for group visits and brief motivational interviewing for individual visits and follow-up phone calls.
  Interventions: Behavioral: Parent education / behavioral counseling
- Usual Care (Placebo Comparator): Parents of children in the control group will receive usual care from their primary care provider as well as a copy of the NIH We Can! Parent Handbook.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Parent education / behavioral counseling — Providers and study personnel will be trained in the use of the NIH We Can! curriculum for group visits and brief motivational interviewing for individual visits and follow-up phone calls. Training will be conducted by the PI and Co-Investigators using a combination of online, self-study, and face-to-face formats totally at least/approximately 8 hours. At least one project team member will attend each group visit. Specifically, the American Academy of Pediatrics 15-minute Obesity Prevention Protocol will be utilized during individual visits. The intervention is designed to take place over a period of 10-12 weeks in the primary care office.
  Arms: Parent education / behavioral counseling
Behavioral: Usual Care — Parents of children in the control group will receive usual care from their primary care provider as well as a copy of the NIH We Can! Parent Handbook.
  Arms: Usual Care

SUMMARY:
Child overweight has become one of today's most important public health concerns. Engaged and skilled parenting that models, values, and encourages healthy eating habits and a physically active lifestyle can play a key role in childhood overweight prevention and reduction. Primary care providers are well positioned to intervene with children and their parents, but face many barriers in addressing child overweight. A child overweight treatment approach is proposed for the primary care setting to facilitate parents' active involvement and self-efficacy in promoting healthy eating habits and physical activity for their children. We will test the following hypotheses: Hypothesis I (primary hypothesis): Children assigned to the intervention group will improve more in weight status (measured by BMI percentile) than children in the control group. Hypothesis II: Primary care providers assigned to the intervention group will improve more in their competence in addressing child overweight than the providers in the control group. Hypothesis III: After the intervention, parents in the intervention group will have more involvement and self-efficacy in promoting healthy weight for their children than parents in the control group. Hypothesis IV: Compared to the control group, the intervention group will improve more in family diet and eating, physical activity behaviors, as well as parental attitude and beliefs. Eighty children five to eleven years old who are overweight or obese will be recruited from two pediatric and two family practice clinics in southern Appalachia. Children will be randomly assigned to intervention and control groups based on clinic affiliation. Parents of children in the intervention group will participate in four clinic-based group sessions using the NIH We Can! curriculum moderated by a trained clinic provider, two individual brief motivational interviewing visits with their clinic provider, and four follow-up phone calls with the project coordinator or registered dietician. Parenting behaviors and attitudes, and family eating and activity habits, and children's weight status will be assessed at baseline, at the completion of the intervention, and at six months after the intervention. Changes in the assessments will be compared between treatment and control groups. Changes in provider and parent attitudes and perceptions about this treatment approach,adherence to the program, and estimates of associated time will be measured.

DETAILED DESCRIPTION:
Specific aims of this project are: 1) to establish a primary care based and parent-mediated childhood overweight intervention program based on the Chronic Care Model in the primary care setting, 2) to explore the efficacy of this intervention in improving the weight status of children, 3) to examine the acceptability and feasibility of the approach among primary care providers and parents. Clinic providers and study personnel will be trained in the use of brief motivational interviewing (brief MI) for the visits and phone calls. The American Academy of Pediatrics 15-Minute Obesity Prevention Protocol will be used for individual visits while the NIH We Can! curriculum and materials will be used for group visits. Parents in the control group will receive the We Can! Parent Handbook and usual care. The intervention is designed to facilitate efficient communication of advice about behavior change, nutrition, and physical activity to parents. Partnership of primary care providers with parents and use of brief intervention techniques and group visits can be a practical approach. If proven to be effective, this approach can serve as an exportable model to other primary care practices and will reach a large proportion of the population and have far-reaching effects.

ELIGIBILITY:
Inclusion Criteria:

* BMI >= 85th percentile
* age 5-11 years
* one parent or other primary care giver agrees to participate in the study

Exclusion Criteria:

* current participation in another weight management program by child or parent/caregiver
* presence of a diagnosed psychiatric/psychological disorder in the parent or child
* presence of an underlying condition affecting weight status
* current dietary or physical activity limitations
* parents who do not have phone accessibility

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2009-09; Primary Completion 2010-11 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
child body mass index percentile | 6 months

SECONDARY OUTCOMES:
Parent report of knowledge, attitudes, perceptions, intentions, and behaviors related to eating and physical activity | 6 months

OTHER OUTCOMES:
Health care provider knowledge, attitudes, and practices related to child obesity management | 6-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen E Schetzina, MD, MPH, Principal Investigator — East Tennessee State University
Locations (1):
- East Tennessee State University, Johnson City, Tennessee, United States

REFERENCES:
- [Background] Dalton WT 3rd, Schetzina KE, Holt N, Fulton-Robinson H, Ho AL, Tudiver F, McBee MT, Wu T. Parent-Led Activity and Nutrition (PLAN) for healthy living: design and methods. Contemp Clin Trials. 2011 Nov;32(6):882-92. doi: 10.1016/j.cct.2011.07.004. Epub 2011 Jul 18. PMID 21777701
- [Result] Holt N, Schetzina KE, Dalton WT 3rd, Tudiver F, Fulton-Robinson H, Wu T. Primary care practice addressing child overweight and obesity: a survey of primary care physicians at four clinics in southern Appalachia. South Med J. 2011 Jan;104(1):14-9. doi: 10.1097/SMJ.0b013e3181fc968a. PMID 21119559